CLINICAL TRIAL: NCT03610516
Title: A Randomized, Placebo-controlled, Patient and Investigator Blinded, Study Investigating the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Multiple Doses of CFZ533 in Patients With Moderately Active Proliferative Lupus Nephritis
Brief Title: Safety, Pharmacokinetics and Preliminary Efficacy Study of CFZ533 in Patients With Lupus Nephritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCFZ533X2202
Record Dates: First submitted 2018-06-01; First posted 2018-08-01 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Lupus Nephritis
Keywords: anti-CD40; CFZ533; moderately active lupus nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — iscalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CFZ533 (Experimental): Investigational drug CFZ533 will be administred as multiple doses
  Interventions: Drug: CFZ533
- Placebo (Placebo Comparator): Investigational drug matching placebo will be administered as multiple doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CFZ533 — Multiple doses of 10 mg/kg CFZ533 intravenous (IV) infusion. CFZ533 was administered every 4 weeks (Q4W; from Day 1 to Day 141), plus an additional dose of 10 mg/kg IV at Day 15, resulting in a Q2W loading regimen up to the third dose on Day 29.
  Arms: CFZ533
Drug: Placebo — multiple doses of placebo intravenous infusion
  Arms: Placebo

SUMMARY:
This study was to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary therapeutic efficacy of multiple doses of CFZ533 anti-CD40 monoclonal antibody in patients with moderately active lupus nephritis.

DETAILED DESCRIPTION:
This was a randomized, subject and investigator blind, placebo controlled multicenter study with multiple doses of CFZ533 administered by 1-hour intravenous infusion over a 24 week treatment period, as compared to matched placebo infusion. The treatment period was followed by a 24-week safety follow-up period.The duration of the study (including the screening period) for each patient was approximately 53 weeks. The investigational drug or placebo was administered on top of standard of care therapy for lupus nephritis.

Patients were screened within 29 days of the first study drug infusion. Eligibility was confirmed at the baseline visit within one week before the first dose. Eligible patients were assigned a randomization number and receive the intravenous infusion within 3 days of baseline visit.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women with systemic lupus erythematosus (SLE) aged ≥ 18 years and ≤ 75 years at screening, fulfilling at least 4 out of 11 criteria for SLE as defined by the American College of Rheumatology (Tan at al 1982, revised by Hochberg 1997)
* Subjects must have a body mass index (BMI) within the range of 18 - 40 kg/m2 at screening visit
* Histological diagnosis of proliferative lupus nephritis World Health Organization (WHO) ISN/RPS (Weening et al 2004) Class III or IV within 5 years of screening
* Presence of antinuclear autoantibody (ANA titer ≥ 1:80) at screening
* Morning UPCR ≥ 0.5 at screening visit and baseline visit
* At least one of the following:

  1. low complement level (C3 ˂ 0.9 g/L) or (C4 ˂ 0.1 g/L), and/or
  2. elevated anti-dsDNA (≥ 30 IU/mL), and/or
  3. urine sediment consistent with active proliferative LN such as presence of cellular (granular or red blood cell) casts or hematuria ( ˃5 red blood cells per high power field) if other causes such as menstrual bleeding are excluded
* Patient must have sufficient kidney function as estimated by eGFR ˃ 30mL/min/1.73 m2 at screening and baseline visits (Levey et al 2009)
* Patient must have active disease as defined by proteinuria and additional symptoms as above despite standard of care therapy for LN as considered appropriate by the treating physician (e.g., corticosteroids and/or immunosuppressive or immunomodulatory treatments such as mycophenolate, azathioprine, methotrexate or hydroxychloroquine). For guidance, see published guidelines such as Bertsias et all 2012 and Hahn et al 2012.
* Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) must use highly effective methods of contraception during dosing and until study completion.

Key Exclusion Criteria:

* Any glomerulonephritis other than WHO Class III or IV lupus nephritis. Patients with proliferative nephritis (Class III or IV) who, in addition, have overlapping histological signs for other glomerulonephritis, e.g., Class V, are eligible at the investigator´s discretion.
* Hypoalbuminemia (serum albumin of less than 2.0 g/dL)
* Patients who have received:

  1. oral or i.v. cyclophosphamide within 3 months prior to randomization
  2. i.v. corticosteroid bolus (dose ˃ 1 mg/kg) within 3 months prior to randomization
  3. rituximab or other B cell depleting agent within 12 months. for patients who received such treatment earlier, B cell count should be within normal ranges prior to randomization
  4. belimumab within 6 months prior to randomization
  5. any other biologic drug or an investigational drug within one months or five times the half-life, whichever is longer prior to randomization
  6. any calcineurin inhibitor (e.g., tacrolimus or cyclosporin A) within 3 months prior to randomization
* Patients who are at significant risk for the thromboembolic events based on the following:

  1. history of either thrombosis or 3 or more spontaneous abortions
  2. presence of lupus anticoagulant or prolonged activated partial thromboplastin time (aPTT) and no prophylactic treatment with aspirin or anticoagulants as per local standard of care
* Have had signs or symptoms of a clinically significant systemic viral, bacterial or fungal infection within 30 days prior to randomization
* Live vaccines within 4 weeks of the first study drug infusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- Argentina (2):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Córdoba
- China (5):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Mainz, Germany
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Debrecen, Hungary
- Russia (3):
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- South Korea (2):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Tunis, Tunisia
- Novartis Investigative Site, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Shen N, Weinmann-Menke J, Malvar A, Serra-Roma A, Weiss M, Danekula R, Sips C, Rohr J, Felten R, Gergely P, Shisha T. Efficacy, pharmacokinetics and safety of iscalimab (CFZ533) in patients with proliferative lupus nephritis: a randomised, double-blind, placebo-controlled, phase II study. RMD Open. 2025 Aug 14;11(3):e005557. doi: 10.1136/rmdopen-2025-005557. PMID 40813108
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2171

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 21 investigative sites in 10 countries.
Pre-assignment Details: There was a screening period within 29 days to assess participants eligibility. After last dose of study treatment patients could enter the post-treatment follow-up.
Groups:
- CFZ533 10 mg/kg i.v.: CFZ533 10 mg/kg i.v. dose on Day 1, 15, 29, 57, 85, 113, and 141
- Placebo i.v.: Placebo i.v. dose on Day 1, 15, 29, 57, 85, 113, and 141
Period: Treatment Epoch
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Started | 39 | 18
Completed | 21 | 10
Not Completed | 18 | 8
Not completed — Adverse Event | 3 | 1
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — No longer requires treatment | 1 | 0
Not completed — Non-Compliance with study treatment | 1 | 0
Not completed — Physician Decision | 8 | 5
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Period: Post-Treatment Follow-up
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Started | 34 | 16
Completed | 32 | 16
Not Completed | 2 | 0
Not completed — Subject/Guardian Decision | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v. | Total
Number analyzed (Participants) | 39 | 18 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (9.20) | 36.4 (9.15) | 34.8 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 17 | 47
  Male | 9 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 7 | 23
  Asian | 23 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness), AEs led to study treatment discontinuation, SAEs and SAEs led to study treatment discontinuation.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 49 weeks.
Population: The safety analysis set included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 39 | 18
Participants
  Adverse Events | 33 | 18
  Serious Adverse Events | 6 | 3
  AEs leading to discontinuation of study treatment | 3 | 1
  SAEs leading to discontinuation of study treatment | 0 | 0

2. Primary Outcome: Ratio to Baseline in Urinary Protein Creatinine Ratio (UPCR)
Description: A urine protein creatinine ratio (UPCR) test is a urine test. It measures the levels of protein and creatinine in urine. UPCR was assessed using the first morning void if available at a visit otherwise using the clinic spot sample, and was expressed as protein/creatinine (mg/mmol). High UPCR values can be a sign of kidney disease. An UPCR ratio to baseline <1 indicates improvement from baseline.
Time Frame: Baseline, Day 169
Population: Participants in the pharmacodynamics (PD) analysis set with an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio to baseline in UPCR
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 20 | 10
ratio to baseline in UPCR | 0.369 [0.234 to 0.582] | 0.637 [0.338 to 1.202]
Statistical Analysis 1: Comparison: CFZ533 10 mg/kg i.v. vs Placebo i.v; Test type: Other — A repeated measures mixed model was fitted with factors for treatment group (CFZ533 or placebo) and visit; p = 0.0788, Repeated measures Mixed Model — one-sided p-value; Ratio of geometric means CFZ533/placebo = 0.579, 95% CI 2-sided [0.267 to 1.256]

3. Secondary Outcome: Ratio to Baseline for Urine Protein Creatinine Ratio (UPCR)
Description: as for outcome 2
Time Frame: Day 197, Day 225, Day 253, Day 281, Day 309, Day 337 (End of Study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio to baseline in UPCR
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 35 | 16
ratio to baseline in UPCR
  Day 197 | 0.532 (0.4160) | 0.985 (0.9045)
  Day 225: number analyzed (Participants) | 32 | 16
  Day 225 | 0.456 (0.3876) | 1.153 (1.2178)
  Day 253: number analyzed (Participants) | 33 | 14
  Day 253 | 0.648 (1.3314) | 0.667 (0.3612)
  Day 281: number analyzed (Participants) | 27 | 13
  Day 281 | 0.526 (0.5440) | 0.701 (0.7690)
  Day 309: number analyzed (Participants) | 26 | 12
  Day 309 | 0.580 (0.7175) | 1.101 (1.1337)
  Day 337: number analyzed (Participants) | 20 | 10
  Day 337 | 0.640 (0.7446) | 0.735 (0.5323)

4. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) of CFZ533
Description: Pharmacokinetic parameters were directly derived from the PK concentration data using non-compartmental analysis. AUClast is the area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (tlast) of free CFZ533.
Time Frame: Day 141: pre dose and 1 hour post dose
Population: Participants in the Pharmacokinetic (PK) analysis set with an available value for the outcome measure. The (PK) analysis set included all subjects with at least one available valid PK concentration measurement, who received any study drug and with no protocol deviations that impact on PK data. The PK analysis set is only applicable to the CFZ533 arm.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | CFZ533 10 mg/kg i.v.
Number analyzed (Participants) | 11
day*ug/mL | 7250 (1800)

5. Secondary Outcome: Pre-dose Trough Concentration (Ctrough) of CFZ533
Description: Pharmacokinetic parameters were directly derived from the PK concentration data using non-compartmental analysis. Ctrough is the observed plasma concentration that is just prior to the beginning of, or at the end of a dosing interval.
Time Frame: Pre-dose at: Day 1, Day 15, Day 29, Day 57, Day 85, Day 113 and Day 141
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CFZ533 10 mg/kg i.v.
Number analyzed (Participants) | 33
ug/mL
  Day 1 | 0 (0)
  Day 15: number analyzed (Participants) | 14
  Day 15 | 49.8 (37.0)
  Day 29: number analyzed (Participants) | 30
  Day 29 | 64.1 (31.6)
  Day 57: number analyzed (Participants) | 15
  Day 57 | 34.5 (21.7)
  Day 85: number analyzed (Participants) | 25
  Day 85 | 33.2 (25.0)
  Day 113: number analyzed (Participants) | 26
  Day 113 | 32.7 (26.3)
  Day 141: number analyzed (Participants) | 21
  Day 141 | 34.1 (26.6)

6. Secondary Outcome: The Observed Maximum Plasma Concentration Following CFZ533 Administration at Steady State (Cmax,ss)
Description: Pharmacokinetic parameters were directly derived from the PK concentration data using non-compartmental analysis. Cmax,ss is the observed maximum plasma concentration following CFZ533 administration at steady state [mass/volume].
Time Frame: Day 141: pre dose and 1 hour post dose
Population: Participants in the Pharmacokinetic (PK) analysis set with an available value for the outcome measure. The PK analysis set included all subjects with at least one available valid PK concentration measurement, who received any study drug and with no protocol deviations that impact on PK data. The PK analysis set is only applicable to the CFZ533 arm.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CFZ533 10 mg/kg i.v.
Number analyzed (Participants) | 20
ug/mL | 263 (81.8)

7. Secondary Outcome: Total Soluble CD40 Plasma Concentrations
Description: Total soluble CD40 concentrations in plasma. An increase in soluble CD40 concentrations is considered a marker for CFZ533 target engagement. This endpoint is only applicable to the CFZ533 arm.
Time Frame: Day 1, Day 15, Day 29, Day 57, Day 113, Day 169, Day 225, Day 281, Day 337 (End of Study)
Population: Participants in the Pharmacodynamics (PD) analysis set who received CFZ533 and had an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CFZ533 10 mg/kg i.v.
Number analyzed (Participants) | 30
ng/mL
  Day 1 | 0.2723 (0.22222)
  Day 15: number analyzed (Participants) | 16
  Day 15 | 78.7375 (20.58802)
  Day 29: number analyzed (Participants) | 28
  Day 29 | 90.4286 (23.86165)
  Day 57: number analyzed (Participants) | 14
  Day 57 | 127.6214 (26.11617)
  Day 113: number analyzed (Participants) | 24
  Day 113 | 109.2672 (50.19834)
  Day 169: number analyzed (Participants) | 7
  Day 169 | 158.5714 (22.24753)
  Day 225: number analyzed (Participants) | 16
  Day 225 | 8.3406 (17.77703)
  Day 281: number analyzed (Participants) | 15
  Day 281 | 0.7981 (0.32464)
  Day 337 (End of Study): number analyzed (Participants) | 13
  Day 337 (End of Study) | 0.5331 (0.30080)

8. Secondary Outcome: Number of Participants With Anti-CFZ533 Antibodies
Description: To evaluate the immunogenicity of CFZ533 via the quasi-quantitative analysis of anti-CFZ533 antibodies.
Time Frame: Day 1, Day 15, Day 29, Day 57, Day 113, Day 169, Day 225, Day 281, Day 337 (End of study)
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 33 | 16
Participants
  Day 1-Negative: number analyzed (Participants) | 33 | 13
  Day 1-Negative | 32 | 13
  Day 1-Positive: number analyzed (Participants) | 33 | 13
  Day 1-Positive | 1 | 0
  Day 15-Negative: number analyzed (Participants) | 17 | 8
  Day 15-Negative | 17 | 8
  Day 15-Positive: number analyzed (Participants) | 17 | 8
  Day 15-Positive | 0 | 0
  Day 29-Negative | 33 | 16
  Day 29-Positive | 0 | 0
  Day 57-Negative: number analyzed (Participants) | 17 | 8
  Day 57-Negative | 17 | 8
  Day 57-Positive: number analyzed (Participants) | 17 | 8
  Day 57-Positive | 0 | 0
  Day 113-Negative: number analyzed (Participants) | 32 | 15
  Day 113-Negative | 32 | 15
  Day 113-Positive: number analyzed (Participants) | 32 | 15
  Day 113-Positive | 0 | 0
  Day 169-Negative: number analyzed (Participants) | 14 | 8
  Day 169-Negative | 14 | 8
  Day 169-Positive: number analyzed (Participants) | 14 | 8
  Day 169-Positive | 0 | 0
  Day 225-Negative: number analyzed (Participants) | 26 | 13
  Day 225-Negative | 25 | 13
  Day 225-Positive: number analyzed (Participants) | 26 | 13
  Day 225-Positive | 1 | 0
  Day 281-Negative: number analyzed (Participants) | 24 | 13
  Day 281-Negative | 23 | 13
  Day 281-Positive: number analyzed (Participants) | 24 | 13
  Day 281-Positive | 1 | 0
  Day 337-Negative (EOS): number analyzed (Participants) | 13 | 8
  Day 337-Negative (EOS) | 12 | 8
  Day 337-Positive (EOS): number analyzed (Participants) | 13 | 8
  Day 337-Positive (EOS) | 1 | 0

9. Secondary Outcome: Hematuria Casts- Urine White Blood Cell Casts
Description: Urine was tested using a dipstick. If the dipstick result was positive for protein, nitrite, leucocytes and/or blood, a microscopic analysis of white blood cells (WBC), red blood cells (RBC) and casts was performed. Hematuria is the presence of blood in the urine. Hematuria casts were assessed by microscopic urinalysis and classified as granular casts and WBC casts. Only in the event of a positive result, these samples were submitted to reflex testing microscopic analysis for counting of casts which resulted in a numeric value related to the number of respective casts presented in the urine.
Time Frame: Baseline, Day 1 (Pre dose), and Day 309
Population: Participants in the pharmacodynamics (PD) analysis set with a microscopic urinalysis and an available value for the outcome measure at baseline and the corresponding time point. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: number of casts per low power field
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 37 | 18
number of casts per low power field
  Baseline: number analyzed (Participants) | 1 | 0
  Baseline | 2 |
  Day 1: number analyzed (Participants) | 1 | 0
  Day 1 | 2 |
  Day 309: number analyzed (Participants) | 1 | 0
  Day 309 | 4 |

10. Secondary Outcome: Hematuria Casts- Casts Granular
Description: as for outcome 9
Time Frame: Day 1 (Pre dose), Day 15 (Pre dose), Day 29 (Pre dose), Day 253, and Day 337 (end of study)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of casts per low power field
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 37 | 18
number of casts per low power field
  Day 1: number analyzed (Participants) | 1 | 0
  Day 1 | 3 |
  Day 15: number analyzed (Participants) | 2 | 0
  Day 15 | 2.5 (0.71) |
  Day 29: number analyzed (Participants) | 0 | 2
  Day 29 |  | 3 (1.41)
  Day 253: number analyzed (Participants) | 1 | 0
  Day 253 | 14.0 |
  Day 337 (End of Study): number analyzed (Participants) | 2 | 0
  Day 337 (End of Study) | 5 (2.83) |

11. Secondary Outcome: Change From Baseline in Urine Hyaline Casts
Description: Urine was tested using a dipstick. If the dipstick result was positive for protein, nitrite, leucocytes and/or blood, a microscopic analysis of white blood cells (WBC), red blood cells (RBC) and casts was performed.
  Urine hyaline casts were assessed by microscopic urinalysis.
Time Frame: Baseline, Day 1 (Pre dose), Day 15 (Pre dose), Day 29 (Pre dose), Day 57 (Pre dose), Day 85 (Pre dose), Day 113 (Pre dose), Day 141 (Pre dose), Day 169, Day 197, Day 225, Day 253, Day 281, Day 309 and Day 337 (end of study)
Population: Participants in the pharmacodynamics (PD) analysis set with a microscopic urinalysis and an available value for the outcome measure at baseline and the corresponding time point. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. The participants analyzed are the ones with available value for the outcome measure at baseline and the corresponding time point.
Measure: Mean (Standard Deviation); unit: number of casts per low power field
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 37 | 18
number of casts per low power field
  Day 1: number analyzed (Participants) | 0 | 0
  Day 15: number analyzed (Participants) | 4 | 3
  Day 15 | 8.3 (15.88) | 3.7 (3.51)
  Day 29: number analyzed (Participants) | 4 | 4
  Day 29 | 2.8 (4.99) | 5.0 (2.16)
  Day 57: number analyzed (Participants) | 3 | 2
  Day 57 | -5.0 (3.61) | 1.0 (1.41)
  Day 85: number analyzed (Participants) | 2 | 1
  Day 85 | 0.5 (2.12) | -4.0
  Day 113: number analyzed (Participants) | 0 | 3
  Day 113 |  | 18.0 (28.58)
  Day 141: number analyzed (Participants) | 0 | 2
  Day 141 |  | -4.5 (6.36)
  Day 169: number analyzed (Participants) | 1 | 1
  Day 169 | 0.0 | 0.0
  Day 197: number analyzed (Participants) | 3 | 3
  Day 197 | -1.0 (2.65) | 2.7 (9.02)
  Day 225: number analyzed (Participants) | 1 | 1
  Day 225 | 2.0 | 0.0
  Day 253: number analyzed (Participants) | 0 | 2
  Day 253 |  | -0.5 (4.95)
  Day 281: number analyzed (Participants) | 1 | 2
  Day 281 | 0.0 | -1.5 (4.95)
  Day 309: number analyzed (Participants) | 3 | 1
  Day 309 | 1.7 (1.15) | -4.0
  Day 337 (EOS): number analyzed (Participants) | 0 | 2
  Day 337 (EOS) |  | 0.5 (0.71)

12. Secondary Outcome: Number of Participants Who Fulfil the Criteria for Complete Renal Remission (CRR)
Description: The criteria for CRR were defined as:
  1. Urinary protein creatinine ratio (UPCR) ≤ 0.2 mg/mg
  2. Estimated glomerular filtration rate (eGFR) ≤ 25% of Baseline
  3. Normal urine sediment.
  If the UPCR from the first morning void sample was not available, then the UPCR from the corresponding spot sample taken at the investigator site was used in the derivation of complete renal remission.
Time Frame: Baseline, up to Day 169
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 37 | 18
Participants | 13 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 49 weeks.
Groups:
- CCFZ533 10mg/kg: CFZ533 10 mg/kg i.v. dose on Day 1, 15, 29, 57, 85, 113, and 141
- All Patients: All patients
Arm/Group | CCFZ533 10mg/kg | Placebo i.v. | All Patients
All-Cause Mortality (participants affected / at risk) | 2/39 | 0/18 | 2/57
Serious Adverse Events (participants affected / at risk) | 6/39 | 3/18 | 9/57
Other Adverse Events (participants affected / at risk) | 32/39 | 18/18 | 50/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CCFZ533 10mg/kg (N=39) | Placebo i.v. (N=18) | All Patients (N=57)
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CCFZ533 10mg/kg (N=39) | Placebo i.v. (N=18) | All Patients (N=57)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Corneal erosion (Eye disorders) | 0 | 1 | 1
Eyelid bleeding (Eye disorders) | 1 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 2 | 0 | 2
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 2 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1 | 2
COVID-19 (Infections and infestations) | 5 | 3 | 8
Conjunctivitis (Infections and infestations) | 1 | 1 | 2
Cystitis (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 2 | 2
Herpes zoster (Infections and infestations) | 3 | 1 | 4
Influenza (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0 | 4
Peri-implantitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0 | 1
Pyuria (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 1
Tinea cruris (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 2 | 9
Urinary tract infection (Infections and infestations) | 2 | 3 | 5
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood immunoglobulin G decreased (Investigations) | 1 | 0 | 1
Blood immunoglobulin M decreased (Investigations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 2 | 0 | 2
Neutrophil count increased (Investigations) | 3 | 0 | 3
Protein urine present (Investigations) | 0 | 1 | 1
Red blood cell sedimentation rate increased (Investigations) | 1 | 1 | 2
Systemic lupus erythematosus disease activity index abnormal (Investigations) | 1 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0 | 1
Urine protein/creatinine ratio increased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 3
Occipital neuralgia (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 2
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Lupus nephritis (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT03610516/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT03610516/SAP_001.pdf